CLINICAL TRIAL: NCT06699823
Title: Cultural Adaptation and Validation of the Greek Version of the Postoperative Quality of Recovery Score 15 (QoR-15Gr)
Brief Title: Validation of the Greek Postoperative Quality of Recovery Score 15
Acronym: (QoR-15Gr)
Status: Not yet recruiting | Type: Observational
Sponsor: IASO Thessalias (Other)
Responsible Party: Principal Investigator, DESPOINA LIOTIRI, Anesthesiologist, IASO Thessalias
Other Study IDs: 785
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Recovery; Quality of Recovery From Anaesthesia; PROMs; Validation Study; Cultural Adaptation
Keywords: quality of recovery; patient reported outcomes; QoR-15; validation; cultural adaptation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Greek version of QoR-15 — Greek version of QoR-15

SUMMARY:
The goal of this observational study is to translate a patient questionnaire about recovery after an operation into Greek and assess how accurate, reliable, acceptable, and feasible this Greek version is.

DETAILED DESCRIPTION:
This study aims to culturally adapt and validate a Greek version of the Quality of Recovery - 15 (QoR-15), referred to as the QoR-15Gr, for Greek-speaking surgical patients. The investigators hypothesize that the QoR-15Gr will demonstrate psychometric properties comparable to the original English version.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Scheduled elective general surgery under general anesthesia

Exclusion Criteria:

* Emergency surgery
* Poor Greek comprehension
* Inability to give consent
* A psychiatric or neurological condition that precludes cooperation
* Known history of alcohol or drug dependence
* Life-threatening postoperative complications
* Postoperative admission to ITU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will take place in IASO Thessalias General Hospital (the largest private general hospital in the region of Thessaly in Greece).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Translation and cultural adaptation of the Greek version of the postoperative quality of recovery score 15 (QoR-15Gr) | From enrollment until 20 first patient have been enrolled
  The QoR-15 consists of 15 questions and the patients are asked to rate various aspects of their postoperative recovery from 0 to 10. Minimum score is 0 and corresponds to the worst score. Maximum score is 150 and corresponds to optimal recovery.
  Translation into Greek and pilot test will be performed.
Psychometric properties of postoperative quality of recovery 15 (QoR-15Gr) will be assessed by evaluating validity (convergent, construct, and discriminant), reliability (internal consistency and repeatability), and responsiveness. | From enrollment until 150 patients have been enrolled
Acceptability and feasibility of the postoperative quality of recovery 15 (QoR-15Gr) will be assessed by measuring patient recruitment rate as well as successful recruitment rate. | From enrollment until 150 patients have been enrolled

CONTACTS AND LOCATIONS:
Overall Officials: DESPOINA LIOTIRI, ANAESTHESIOLOGIST, Principal Investigator — IASO THESSALIAS GENERAL HOSPITAL; DIMITRIOS ZACHAROULIS, PROFESSOR OF SURGERY, Study Chair — University of Thessaly
Locations (1):
- IASO Thessalias General Hospital, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No